CLINICAL TRIAL: NCT05612399
Title: Precision Perioperative Methadone Use in Adult Cardiac Surgical Patients to Reduce Opioid Use Adverse Effects While Improving Analgesia and Outcomes
Brief Title: Precision Analgesia for Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Kathirvel Subramaniam (Other)
Responsible Party: Sponsor-Investigator, Kathirvel Subramaniam, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY22060101
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-04

CONDITIONS: Analgesia; Cardiac Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One Pharmacogenetic (PG) blood sample collection of 1-3mL obtained prior to surgery. Genotyping will include ABCB1, CYP2B6, OPRM1, FAAH, CYP2D6, ORM1, and CYP3A4. Other relevant exploratory genes in custom gene panel will include ADRB2, GCH1, TRPA1, COMT, and DRD2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The proposed research is an important extension of an ongoing perioperative personalized analgesia and intravenous opioid pharmacogenetic research. This research focuses on two of the most commonly used oral opioid analgesics, oxycodone, and methadone in elderly adults undergoing cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery patients often experience significant acute postoperative pain, and untreated or undertreated pain has consequences. Each year, 900,000 painful cardiac surgeries occur in the US alone. Pain associated with cardiac surgery results from surgical incision, sternal retraction, internal mammary artery harvesting, saphenous vein removal, placement of mediastinal and chest drains, sternal wires, and release of pro-inflammatory mediators after tissue injury. One study reported that 49%, 62%, and 78% of patients reported severe pain at rest, movement, and coughing, respectively after coronary artery bypass surgery (CABG). Another study showed that 61.4% of patients undergoing cardiac surgery reported moderate to severe pain. Inadequate pain treatment is common in cardiac surgery due to health care providers' fears of causing cardiorespiratory compromise. Poor pain control can trigger sympathoadrenal responses leading to cardiac arrhythmias and myocardial ischemia, restrict mobility to cause venous thrombosis, impair clearance of secretions leading to pulmonary complications such as atelectasis and pneumonia, decrease patient satisfaction and predispose to the development of chronic, persistent surgical pain (CPSP).

Improving clinical practice by shifting paradigms: Our research is transformative and will evolve current reactive clinical practice towards proactive precision methods based on genetic risks for surgical pain and ORADE in elderly vulnerable population. This is the first effort to move in the direction of personalizing perioperative opioid use with precise dosing to improve safety and efficacy in cardiac surgery. Preoperative genotyping-based clinical decisions are expected to support clinical implementation in real-world settings. Importantly, investigators will be able to reach beyond the current best-in-class outcomes with precision multi-dose methadone analgesia based on proactive genetic risk identification to maximize safety and efficacy of opioids in all cardiac surgical patients and positively impact socio-economic outcomes in the future. By addressing these critical barriers, this research will help physicians identify patients at risk and improve the safety and efficacy of opioids and surgical pain management while preventing OD, misuse, overdose, and deaths.

ELIGIBILITY:
Inclusion Criteria:

* Elderly cardiac surgical patients over 60 years of age

Exclusion Criteria:

* Methadone allergy
* Morbid obesity (BMI >40kg/cm2)
* Severe sleep apnea
* Severe pulmonary disease requiring oxygen therapy
* Preoperative mechanical circulatory support
* Emergency surgery
* Liver disease (liver enzymes more than two times normal)
* End-stage renal disease requiring dialysis
* Serum creatinine more than 2.0mg

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly cardiac surgical patients over 60 years of age Both genders are included All races and ethnic groups undergoing elective open cardiac surgery through midline sternotomy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine Genetic Factors - Opioid Related Adverse Events (RD) | Immediately post-surgery during hospital stay
  Respiratory depression will be measured with binary yes/no responses obtained either via self-report from the patient or reported by the clinical care staff.
Determine Genetic Factors - Opioid Related Adverse Events (PONV) | Immediately post-surgery during hospital stay
  Post-operative nausea and vomiting will be measured with binary yes/no responses obtained either via self-report from the patient or reported by the clinical care staff.
Determine Genetic Factors - Opioid Related Adverse Events (Excessive Sedation) | Immediately post-surgery during hospital stay
  Excessive sedation will be measured with binary yes/no responses obtained either via self-report from the patient or reported by the clinical care staff.
Determine Genetic Factors - Uncontrolled severe pain | Immediately post-surgery during hospital stay
  We postulate that specific CYP2B6, ABCB1, OPRM1, FAAH, and ORM1 genetic variants identify patients at risk for poor pain relief and ORADE with methadone in the immediate post-surgical period. Pain will be measured by the Numerical Rating Scale (NRS) in which 0 = no pain at all and 10 = worst pain imaginable. This will be self-reported responses by the patient.

SECONDARY OUTCOMES:
Opioid use post-operatively | Post-operative Day 5 to 6-months post-operative
  Opioid usage will be recorded via SOAPP-R, a 24-item validated opioid assessment. A score of 18 or higher is considered positive.
Patient-Reported Outcomes Measurement Information System | Post-operative Day 5 to 6-months post-operative
  The PROMIS-29 v2.0 will be collected for this outcome measure. The PROMIS survey is scored by the following T-Score Cut Points: 20-55 = better health, 55-60 = mild, 61-69 = moderate, and 71+ = worse health. The general population mean = 50 (SD = 10).
Incidence of Chronic Persistent Surgical Pain (CPSP) | Post-operative Day 5 to 6-months post-operative
  CPSP will be obtained via patient-self report as yes/no responses for follow-up assessments. This measure will be reported as mean(SD) for positive CPSP subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Kathirvel Subramaniam, MD, MPH, Principal Investigator — University of Pittsburgh; Amy Monroe, MPH, MBA, Study Director — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States